CLINICAL TRIAL: NCT05544708
Title: Using Grassroots Wellness Coaching to Enhance Reach and Sustainability of Behavioral Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20024014; 1R01DK132373 (NIH)
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: cardiometabolic disease
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Cluster randomized design
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Wellness Ambassadors will undergo training to recruit and deliver a lifestyle intervention to members of their social networks. HCL in the intervention group will deliver the intervention immediately following baseline visits and randomization.
  Interventions: Behavioral: Wellness Engagement Intervention
- Delayed Intervention (No Intervention): Wellness Ambassadors will undergo training to recruit and deliver a lifestyle intervention to members of their social networks. HCL in the delayed intervention group will deliver the intervention after 24 week data collection visits are complete.

INTERVENTIONS:
Behavioral: Wellness Engagement Intervention — Train for, recruit participants into, and lead a 12-week lifestyle intervention delivered via weekly group meetings
  Arms: Intervention

SUMMARY:
African American adults that live in economically disadvantaged areas are at an increased risk for obesity and cardiometabolic disease. The treatment program being tested in this research study aims to address these factors and increase outcomes for the study population. The purpose of this research study is to find out about the feasibility and acceptability of using house chats (HC) as a model for a weight loss program in a real-world, community-based setting.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Resident of Petersburg, VA
* Interested in engaging community members in healthy lifestyle changes (e.g., walking, small changes to eating) and willing to engage in these behaviors her/himself

Exclusion Criteria:

* A diagnosis of type 1 diabetes mellitus.
* Currently being treated for cancer.
* Medical conditions that may increase risk for participating in unsupervised exercise, if medical clearance is not provided
* Hospitalization for depression or other psychiatric disorder within the past 12 months.
* Lifetime history of bipolar disorder or psychotic disorder.
* Currently pregnant or lactating, or planning to become pregnant within the study period.
* Current involvement in a weight loss program or current use of weight loss medication.
* Inability to speak, read and write English.
* Planning to move from the Petersburg area within the study period.
* Does not have sufficient numbers of individuals in their social network from which to recruit for the proposed study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: House Chat Leaders (HCL) | 18 months
  The number of house chat leaders successfully recruited, trained, and retained.
Feasibility: Participants | 18 months
  The average number of participants recruited by the HCLs.
Feasibility: Delivery Model | 12 weeks
  The number of intervention sessions delivered; the number of planned session topics that were covered

SECONDARY OUTCOMES:
Acceptability: Attendance | 12 weeks
  The average number of sessions attended by participants.
Acceptability: Retention | 12 weeks
  The average number of HCL and participants who are retained in the program

CONTACTS AND LOCATIONS:
Overall Officials: Moghboeba Mosavel, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT05544708/ICF_000.pdf